CLINICAL TRIAL: NCT06524037
Title: Relationship Between Metabolic Profiles and Chronic Diseases and Neoplasms
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qin DUAN, clinical professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 20240706
Record Dates: First submitted 2024-07-06; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic disorders are involved in the occurrence and development of a variety of chronic diseases and tumors. There are many common risk factors between chronic diseases and tumors. However, the mechanisms of chronic diseases and tumors caused by metabolic disorders are not completely clear. By observing the relationship between metabolic indexes and chronic diseases and tumors, the investigators intend to explore the possible mechanisms of metabolic status participating in the occurrence and development of chronic diseases and tumors.

DETAILED DESCRIPTION:
Metabolic disorders are involved in the occurrence and development of a variety of chronic diseases and tumors, for example, metabolic diseases (hypertension, diabetes, dyslipidemia, obesity, etc.) can mediate the progression of chronic diseases such as heart failure and ischemic encephalopathy. Obesity can increase the risks of endometrial cancer, esophageal cancer, stomach cancer, etc. There are many common risk factors between chronic diseases and tumors, such as age, sex, smoking, genetics, obesity, unhealthy diet and lack of exercise. However, the mechanisms of chronic diseases and tumors caused by metabolic disorders are not completely clear. By observing the relationship between metabolic indexes and chronic diseases and tumors, the investigators intend to explore the possible mechanisms of metabolic status participating in the occurrence and development of chronic diseases and tumors.

ELIGIBILITY:
Inclusion Criteria:

* adult aged ≥18 years old
* Completed health screening

Exclusion Criteria:

* aged <18 years old
* pregnancy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People undergoing physical examination in the first branch of the First Affiliated Hospital of Chongqing Medical University
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
metabolic disorder | through study completion, an average of 1 year
  The degree of metabolic disorder liking the levels of glycolipids
Chronic disease | through study completion, an average of 1 year
  The occurrence of chronic disease
Tumor | through study completion, an average of 1 year
  The occurrence of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Qin Duan, doctor, Study Director — The First Affiliated Hospital of Chongqing Medical University, Chongqing, China.
Locations (1):
- The First Branch of the Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No